CLINICAL TRIAL: NCT04700852
Title: Efficacy of Puressentiel Protective Nasal Spray on Symptoms and Inflammation in Patients With in Allergic Rhinitis
Brief Title: Efficacy of Puressentiel Protective Nasal Spray in Allergic Rhinitis
Acronym: EPPNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Puressentiel (Industry)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A01877-32
Record Dates: First submitted 2020-11-10; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Allergic Rhinitis Due to Grass Pollen; Allergic Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allergic rhinitis (Experimental): Puressentiel protective nasal spray
  Interventions: Device: Puressentiel protective nasal spray

INTERVENTIONS:
Device: Puressentiel protective nasal spray — provocative nasal test with grass pollen and nasal lavage

SUMMARY:
This study is a proof o concept aiming to determine the efficacy of Puressentiel nasal protective spray (PNPS) in patients with allergic rhinitis.

Cross over study, with a nasal provocative test (NPT) in patients with allergic rhinitis sensitized to grass pollen. A day 0 (first NPT) the following outcomes are recorded: allergic Rhinitis control test (ARCT) and Inspiratory nasal peak flow (INPF) before and 30 min after the NPT. Nasal lavage is performed 30 min after the NPT and 3 cytokines (IL4, IL5 and IL13 are measured by ELISA.

An other NPT is performed at day 30 and the same outcomes measured.

30 min before NPT 2 nasal sprays of PNPS are administered in each nostril in a randomized manner and cross over, the patient being is own control.

The primary outcomes ins the IL4, IL5 and IL13 concentrations in the nasal lavage. ARCT and INPF are the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnostic of allergic rhinitis sensitized to grass pollen for more than one year with or without associated asthma

Exclusion Criteria:

* patients sensitized to a perrianual allergen
* patients with viral infection 4 weeks before inclusion
* patients with severe non controlled asthma
* patients with chronic sinusitis
* pregnancy or breast feeding
* patients with hypersensitivity to essential oil (eucalyptus radie)
* epileptic patient
* patients treated with nasal corticosteroid or anti-histamine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of IL-13 in the nasal lavage will be assessed | measurements at day 1 and day 30
  measurement by ELISA

SECONDARY OUTCOMES:
Change in concentration of IL-5 in the nasal lavage will be assessed | Day1 and Day30
  Measurement by ELISA
Change in concentration of IL-4 in the nasal lavage will be assessed | Day1 and Day 30
  Measurement by ELISA
Change in Nasal Inspiratory Peak Flow will be assessed | Day 1 and Day 30
  Measurement with a peak flow meter
Change in Allergic Rhinitis Control test (ARCT) will be assessed | Day 1 and day 2
  5 questions questionnaire score from 0 to 25 (0 worse score), 25 (best score)

IPD SHARING:
Plan to Share IPD: Undecided